CLINICAL TRIAL: NCT05547789
Title: Assessment Of Diabetic Maculopathy Changes After Phacoemulsification by Using Optical Coherence Tomography
Acronym: Maculopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nermeen Mohammed Ali Hashim, Principal investigator, Assiut University
Other Study IDs: Macular changes after phaco
Record Dates: First submitted 2022-08-31; First posted 2022-09-21 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-09

CONDITIONS: Maculopathy
MeSH Terms: conditions — Macular Degeneration | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group
  Interventions: Drug: non steroidal anti inflammatory drugs
- Control group

INTERVENTIONS:
Drug: non steroidal anti inflammatory drugs — effect of non steroidal anti inflammatory drugs on macular changes
  Other Names: optical coherence tomography
  Groups: Study group

SUMMARY:
Investigators aimed to assess the macular changes with OCT after uncomplicated phacoemulsification surgery in diabetic patients with non proliferative diabetic retinopathy (NPDR) at the time of surgery and the effect of perioperative and postoperative topical NSAIDS on macular changes .

DETAILED DESCRIPTION:
Diabetic patients pose a particular challenge because of the tendency for early formation of cataract in them and propensity to develop macular edema after cataract surgery. Macular edema (ME) is a major cause of vision loss after cataract surgery in patients with diabetes .

Macular edema is a common cause of unfavorable visual outcome after cataract surgery. Clinically significant cystoid macular edema (CSME) has a reported incidence of 1% to 2% after cataract surgery. Diabetes has been associated with an increased incidence of postoperative macular edema. The incidence of macular edema on optical coherence tomography (OCT) was 22% in diabetic eyes undergoing cataract surgery. The macular edema after cataract surgery in diabetic patients could be caused by the cataract surgery or diabetes itself, but it might be hard to differentiate between these two causes .

The level of the preexisting diabetic retinopathy (DR), the presence of clinically significant macular edema (CSME) before the surgery, and duration and regulation of diabetes are all important indicators of postoperative CME . Optical coherence tomography (OCT) has been established as a practical method for examining retinal architecture. OCT, with its noninvasive nature, has been proven to be an indispensable tool for diagnosing retinal pathologies, including cystoid macular edema (CME). Many studies have reported incidences of CME and macular thickness changes, determined by OCT following uneventful cataract surgeries .Nonsteroidal anti-inflammatory drugs (NSAIDS) are widely used and studied by cataract surgeons for varied benefits in the perioperative and postoperative period. Nonsteroidal anti-inflammatory drugs (NSAIDs), a class of medications that inhibit cyclooxygenase (COX) enzymes from producing pro-inflammatory prostaglandins, have multiple indications in the perioperative period including pain control, reducing inflammation, improving intraocular mydriasis, and preventing postoperative cystoid macular edema (CME) .Cataract surgeons often use NSAIDs postoperatively to control patient pain, inflammation, and prevent CME, the most prevalent complication affecting postoperative visual recovery .

ELIGIBILITY:
Inclusion Criteria:

Controlled type 2 non proliferative diabetic retinopathy (NPDR) patients. Immature cataract which does not interfere with ocular imaging.

Exclusion Criteria:

* Patient with dense cataract or vitreous hemorrhage interfering with measurement of central macular thickness Chronic uveitis Any posterior segment pathology that could affect retinal thickness Patient with complicated cataract surgery.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: preoperatively ,Nonsteroidal anti inflammatory drugs was used for prophylaxis before surgery at the postoperative week 1 we gave the same medication to this group
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Macular changes in diabetic patients after phacoemulsification | baseline
  Invgatorsiest aimed to examine the macular changes with OCT after uncomplicated phacoemulsification surgery in diabetic patients with non proliferative diabetic retinopathy (NPDR) at the time of surgery and the effect of perioperative and postoperative topical NSAIDS on macular changes .

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed T. Abd Elmonaiem, Prof, Study Director — Assiut University; Gamal El Dein R. Osman, Ass prof, Study Director — Assiut University; Momen M. Aly, Lecture, Study Director — Assiut University
Locations (2):
- Egypt (2):
  - Assuit University, Asyut
  - Egypt, Asyut

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Furino C, Boscia F, Niro A, D'Addario M, Grassi MO, Saglimbene V, Reibaldi M, Alessio G. DIABETIC MACULAR EDEMA AND CATARACT SURGERY: Phacoemulsification Combined With Dexamethasone Intravitreal Implant Compared With Standard Phacoemulsification. Retina. 2021 May 1;41(5):1102-1109. doi: 10.1097/IAE.0000000000002974. PMID 32897932
- See also: DIABETIC MACULAR EDEMA AND CATARACT SURGERY: Phacoemulsification Combined With Dexamethasone Intravitreal Implant Compared With Standard Phacoemulsification — https://pubmed.ncbi.nlm.nih.gov/32897932/